CLINICAL TRIAL: NCT01277471
Title: Effect of Meal Frequency on Insulin Resistance, Insulin Secretion, and Hepatic Fat Content in Subjects With Type 2 Diabetes
Brief Title: Effect of Meal Frequency on Insulin Resistance in Subjects With Type 2 Diabetes
Acronym: Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Hana Kahleova, Dr., Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3142; NT/11238-4 (Other Grant/Funding Number: Ministry of Health of the Czech Republic, grant NT/11238-4)
Record Dates: First submitted 2011-01-06; First posted 2011-01-17 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: meal frequency; type two diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: 6 and 2 meals/day (Experimental): 6 meals/day for the first 12 weeks followed by 2 meals/day for additional 12 weeks at the same caloric restriction (-500 kcal/day)
  Interventions: Behavioral: Meal frequency (6 meals vs. 2 meals/day)
- Arm B: 2 and 6 meals/day (Active Comparator): 2 meals/day for the first 12 weeks followed by 6 meals/day for additional 12 weeks at the same caloric restriction (-500 kcal/day)
  Interventions: Behavioral: 6 meals/day followed by 2 meals/day

INTERVENTIONS:
Behavioral: Meal frequency (6 meals vs. 2 meals/day) — 6 meals/day for 12 weeks followed by 2 meals/day for 12 weeks at the same caloric restriction (-500 kcal/day)
  Arms: Arm A: 6 and 2 meals/day
Behavioral: 6 meals/day followed by 2 meals/day — 2 meals/day for the first 12 weeks followed by 6 meals/day for additional 12 weeks at the same caloric restriction (-500 kcal/day)
  Arms: Arm B: 2 and 6 meals/day

SUMMARY:
Aims and priorities of the project The purpose of this study is to

1. test the effect of frequency of meals (six vs. two meals daily with the same daily caloric restriction of -500 kcal/day) on insulin sensitivity, insulin secretion, and hepatic fat content.
2. characterize some of the mechanisms of action of different frequencies of meals (amount of visceral fat, hepatic fat content, serum concentrations of adipokines, gut hormones, oxidation stress markers).
3. test the ability of the participants to maintain hypocaloric diet on both regimens when educated and left to prepare their meals alone in comparison with those for whom all meals during the study will be provided.

It will be a randomized, crossover study, where 50 individuals with type 2 diabetes will change in a random order two regimens: six, and two meals a day. Each testing period will take three months.

Glucose and lipid metabolism and its regulation will be thoroughly tested at start, and after each 3-months-period (meal test, hyperinsulinemic isoglycemic clamp, indirect calorimetry, MRI scan of the liver, DXA scan, serum concentration determination of selected adipokines, gut hormones, and oxidation stress markers).

Hypothesis The investigators hypothesize that low plasma insulin levels (as achieved by periods of fasting) will reduce insulin resistance and hepatic lipid content. In contrast, frequent meals (and consequent higher plasma levels of insulin) will predispose to non-alcoholic fatty liver disease and insulin resistance. The investigators further hypothesize that the participants will increase their caloric intake with increased meal frequency (in spite of thorough education) when left to prepare their meals in comparison with those for whom all meals will be provided.

DETAILED DESCRIPTION:
Aims and priorities of the project The purpose of this study is to

1. test the effect of frequency of meals (six vs. two meals daily with the same daily caloric restriction of -500 kcal/day) on insulin sensitivity, insulin secretion, and hepatic fat content.
2. characterize some of the mechanisms of action of different frequencies of meals (amount of visceral fat, hepatic fat content, serum concentrations of adipokines, gut hormones, oxidation stress markers).
3. test the ability of the participants to maintain hypocaloric diet on both regimens when educated and left to prepare their meals alone in comparison with those for whom all meals during the study will be provided.

It will be a randomized, crossover study, where 50 individuals with type 2 diabetes will change in a random order two regimens: six, and two meals a day. Each testing period will take three months.

Glucose and lipid metabolism and its regulation will be thoroughly tested at start, and after each 3-months-period (meal test, hyperinsulinemic isoglycemic clamp, indirect calorimetry, MRI scan of the liver, DXA scan, serum concentration determination of selected adipokines, gut hormones, and oxidation stress markers).

Hypothesis The investigators hypothesize that low plasma insulin levels (as achieved by periods of fasting) will reduce insulin resistance and hepatic lipid content. In contrast, frequent meals (and consequent higher plasma levels of insulin) will predispose to non-alcoholic fatty liver disease and insulin resistance. The investigators further hypothesize that the participants will increase their caloric intake with increased meal frequency (in spite of thorough education) when left to prepare their meals in comparison with those for whom all meals will be provided.

Key words Insulin resistance, meal frequency, type 2 diabetes mellitus, non-alcoholic fatty liver disease, adipokines, gut hormones, oxidative stress Methodology Study design: the investigators will use the design of a randomized, crossover study, where 50 individuals with type 2 diabetes will change in a random order the frequency of their meals: six, and two meals a day. Caloric restriction will be the same (-500 kcal/day). Each testing period will take three months. For one half of the participants all meals during the study will be provided. The other half will be thoroughly educated how to maintain their daily caloric intake during both regimens and they will prepare their meals alone.

Study group: 50 individuals with type 2 diabetes treated by diet only or oral hypoglycemic agents, diabetes duration at least 1 year, both men and women, age 30-65 years, BMI 27-50 kg/m². The subjects will be explained aims, methods and risks of the study and they will sign informed consent (Appendix 1).

Regimens: On the six-meals-per-day-regimen, participants will be asked to divide their total caloric intake into six meals and to eat every two or three hours. On the two-meals-per-day-regimen, they will divide their total caloric intake into two meals: the first meal will be eaten between 6 and 10 a.m., the second one between noon and 4 p.m.

Physical activity: Participants will be asked not to change their exercise habits during the study. Physical activity will be monitored using pedometers and standardized questionnaires: International Physical Activity Questionnaire (IPAQ), and Baecke questionnaire.

Procedures:

At the beginning (week 0), and at the end of every 3 months (week 12, and 24), the following procedures and measurements will be performed at each subject (three times in each subject):

1. Common anthropometric investigations (body weight, BMI, waist and hip circumference), blood samples will be taken for laboratory assessments (common laboratory tests, parameters of glucose and lipid metabolism, chosen adipokines, oxidative stress markers, gut hormones, fatty acid composition in serum phospholipids etc.- see analytic methods).
2. Meal test for glucose tolerance assessment after standard breakfast /baguette Crocodille Cheese Gourmet - 180g, energy 452,8 Kcal/1895,7 kJ, composition: carbohydrates 49,2 g (44,55%), proteins 18,5 g (16,74%), lipids 18,8 g (38,7%), of which saturated 6,8 g, monounsaturated 6,0 g, polyunsaturated 5,0 g/. Blood samples for the assessment of glycemia, C- peptide, immunoreactive insulin (IRI) will be taken in 0, 30, 60, 120 and 180 minutes after breakfast.
3. Hyperinsulinemic (1 mU/kg/min) isoglycemic clamp (HIC) 3 hours long with indirect calorimetry. This method allows exact quantification of insulin resistance and energy substrates utilisation.
4. MRI (magnetic resonance imaging) scan of the liver to measure the hepatic fat content.
5. DXA (Dual energy X-ray absorptiometry) scan to measure total body composition and fat content.
6. Insulin secretion and glucose control will be measured during a one-day-stay in the hospital at the end of each regimen. Blood samples will be taken every three hours during the whole day. Urine will be collected during the whole day to measure microalbuminuria and C-peptide waste.

Analytic methods:

Plasma concentrations of selected adipokines (resistin, adiponectin total, HMW- adiponectin, TNFalfa and leptin) and other cytokines and proteins (FABP) will be measured enzymatically using standard kits (ELISA, Linco, USA). Plasma levels of gut hormones will be measured enzymatically usig standard kits (Milliplex, Millipore, USA). Parameters of lipid peroxidation will be determined according to the levels of TBARS by the reaction with thiobarbituric acid and according to the levels of conjugated dienes.

The level of reduced and oxidised glutathione will be determined using HPLC method with fluorescence detection. Ascorbic acid will be determined spectrophotometric reaction with dinitrophenylhydrazine. Concentrations of a- and g-tocopherol in serum will be determined by reverse-phase high performance liquid chromatography (HPLC) with fluorescence detection according to the modified method of Catignani and Biery. The activity of SOD will be analyzed by the reaction of blocking nitrotethrazolium blue reduction and nitrophormasane formation. Catalase activity measurement is based on the ability of H2O2 to produce with ammonium molybdate the color complex detected spectrophotometrically. The activity of gluthathione peroxidase will be monitored by oxidation velocity of gluthathione by Ellman reagent. Serum glucose will be analysed using the glucose-oxidase method Beckman Analyzer (Beckman Instruments Inc., Fullerton, CA, USA), IRI will be determined by radioimmunoassay using an IMMUNOTECH Insulin IRMA kit (IMMUNOTECH as, Prague, Czech Republic), C-peptide using an IMMUNOTECH C-Peptide IRMA kit (IMMUNOTECH as, Prague, Czech Republic) and glycated hemoglobin will be measured by a Bio-Rad Haemoglobin A1c Column Test (Bio-Rad Laboratories GmbH, Munich, Germany).

Fatty acid pattern in serum phospholipids will be measured after lipids extraction according to Folch and separation of lipid fractions by thin-layer chromatography. The methylesters of fatty acids will be separated by gas chromatography.

Eventual effects of different meal frequency regimens will be evaluated due to chosen gene polymorphisms.

Statistic analysis: Will be done with the use of ANOVA tests, pair and unpair t- tests and other statistic methods using standard statistic programs. Estimate of the number of subjects to be recruited was done using power analysis of repeated measurements via statistic software PASS 2005 (Number Cruncher Statistical Systems, Kaysville, UT, USA). Factors included in this model are interindividual factors (control vs. experimental group), intraindividual factors (individual time stadium in the study) and interaction between factors (divergence degree between time profiles in control and experimental group).

Time frame: December 2010-February 2011 recruitment of the participants March 2011 start of the study Group A: 12 weeks 6 meals/day followed by additional 12 weeks of 2 meal/day Group B: 12 weeks 2 meals/day followed by additional 12 weeks of 6 meal/day September 2011 end of the study

All measurements will be done at start, week 12 and week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes for more than 1 year
2. Treatment of T2D. Oral hypoglycemic agents stable for the last 3 months
3. HbA1c ≥4.2 and ≤10.5% (IFCC)
4. Agek 30-70 years
5. Body Mass Index (kg/m2) between 27 and 50
6. Willingness to follow both different dietary regimens
7. The patient has at least 3 of the symptoms of the metabolic syndrome

Exclusion Criteria:

1. Alcoholism or drug abuse
2. Pregnancy, lactation
3. Nonstable medication for diabetes, hypertension or dyslipidemia in the last 3 months
4. Diagnosis of type 1 diabetes
5. Weight loss or weight gain in the last 3 months (> 5% of the total body weight)
6. Cardiostimulant

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Resistance | Insulin resistance will be measured at weeks 0, 12 and 24. Change from baseline to 12 weeks and from week 12 to week 24 will be assessed.
  Insulin Resistance measured by hyperinsulinemic isoglycemic clamp

SECONDARY OUTCOMES:
hepatic fat content | Hepatic fat content will be measured at weeks 0, 12 and 24. Change from baseline to 12 weeks and from week 12 to week 24 will be assessed.
  hepatic fat content measured by magnetic resonance spectroscopy
Insulin Secretion | Insulin secretion will be measured at weeks 0, 12 and 24. Change from baseline to 12 weeks and from week 12 to week 24 will be assessed.
  Insulin secretion measured by meal test (standard breakfast)
insulin sensitivity | Insulin secretion will be measured at weeks 0, 12 and 24.
  Insulin sensitivity will be measured using the isoglycemic hyperinsulinemic clamp.
Fatty acid composition in serum phospholipids | Weeks 0,12 and 24
  Fatty acid composition in serum phospholipids will be measured by gas liquid chromatography.
Gastrointestinal peptides | Weeks 0, 12 and 24
  Gastrointestinal peptides will be measured in response to a standard breakfast at times 0,30,60,120 and 180.
Oxidative stress markers and AGEs | weeks 0,12 and 24
  Oxidative stress markers and AGEs will be measured in a fasting state.

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikanova, Prof., MD, Study Chair — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Kahleova H, Belinova L, Malinska H, Oliyarnyk O, Trnovska J, Skop V, Kazdova L, Dezortova M, Hajek M, Tura A, Hill M, Pelikanova T. Eating two larger meals a day (breakfast and lunch) is more effective than six smaller meals in a reduced-energy regimen for patients with type 2 diabetes: a randomised crossover study. Diabetologia. 2014 Aug;57(8):1552-60. doi: 10.1007/s00125-014-3253-5. Epub 2014 May 18. PMID 24838678